CLINICAL TRIAL: NCT02771405
Title: Impact of Interferon Free Regimens in Patients With Chronic HCV and Successfully Treated HCC
Acronym: FRI-STC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Hepatology & Tropical Medicine Research Institute (Other Government)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Mohamed Hassany, Hepatology & Gastroenterology Consultant , Director of HCC Unit, National Hepatology & Tropical Medicine Research Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4/2016
Record Dates: First submitted 2016-05-06; First posted 2016-05-13 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Hepatitis C, Chronic; Hepatocellular Carcinoma
Keywords: HCV-HCC-DAAs
MeSH Terms: conditions — Hepatitis C, Chronic; Carcinoma, Hepatocellular | interventions — Sofosbuvir; Ribavirin; Simeprevir; daclatasvir; ledipasvir; ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Sofosbuvir +Ribavirin (Experimental): Sofosbuvir 400 mg/day +ribavirin for 24 weeks
  Interventions: Drug: Sofosbuvir; Drug: Ribavirin
- Sofosbuvir+Simeprevir±Ribavirin (Experimental): Sofosbuvir 400 mg/day +Simeprevir 150 mg/day ± ribavirin for 12 weeks
  Interventions: Drug: Sofosbuvir; Drug: Ribavirin; Drug: Simeprevir
- Sofosbuvir+Daclatasvir±Ribavirin (Experimental): Sofosbuvir 400 mg/day +Daclatasvir 60 mg/day ± ribavirin for 12 weeks
  Interventions: Drug: Sofosbuvir; Drug: Ribavirin; Drug: daclatasvir
- Sofosbuvir+Ledipasvir±Ribavirin (Experimental): Sofosbuvir 400 mg/day +Ledipasvir 90 mg/day ±ribavirin for 12 weeks
  Interventions: Drug: Sofosbuvir; Drug: Ribavirin; Drug: Ledipasvir

INTERVENTIONS:
Drug: Sofosbuvir — Sofosbuvir 400 mg orally once daily
  Other Names: Sovaldi®; GS-7977
Drug: Ribavirin — Ribavirin (RBV) 200 mg tablets administered orally in a divided daily dose (< 75 kg = 1000 mg and ≥ 75 kg = 1200 mg)
  Other Names: Copegus®; Rebetol®
Drug: Simeprevir — Simeprevir 150 mg orally once daily
  Other Names: Olysio®; TMC435
  Arms: Sofosbuvir+Simeprevir±Ribavirin
Drug: daclatasvir — Daclatasvir 60 mg orally once daily
  Other Names: clatazev®; BMS-790052
  Arms: Sofosbuvir+Daclatasvir±Ribavirin
Drug: Ledipasvir — Ledipasvir 90 mg orally once daily
  Other Names: Co-formulated with Sofosbuvir in one tablet (Harvoni ® )
  Arms: Sofosbuvir+Ledipasvir±Ribavirin

SUMMARY:
The study will recruit 150 patients with HCV related HCC ,after HCC treatment the patients will undergo treatment with different regimens of DAAs.

DETAILED DESCRIPTION:
The study will recruit 150 patients with HCV related HCC All the studied patients underwent or will undergo one of the curative interventions for HCC either hepatic resection or thermal ablation .

after 1 month of achievement of laboratory and radiological response to HCC intervention the patient will be treated with one of the interferon free regimens :

1. Sofosbuvir+Ribavirin
2. Sofosbuvir+Simeprevir± Ribavirin
3. Sofosbuvir+ Daclatasvir ± Ribavirin
4. Sofosbuvir+ Ledipasvir ± Ribavirin

the treatment duration will be justified either 12 or 24 weeks after treatment the patient will continue on regular follow up to detect HCV cure or recurrence , HCC cure or recurrence and long term follow up of natural history

ELIGIBILITY:
Inclusion Criteria:

* Age 18-70 years old
* Confirmed HCV viremia by PCR
* CHILD Pugh "A" or "B7,B8"
* Confirmed HCC either by laboratory ,imaging or histopathological criteria
* Underwent or candidate for curative intervention for HCC (BCLC stage 0 ,A)
* Willing to be treated for HCV and signing informed consent

Exclusion Criteria:

* Patients below 18 or above 70 years old
* patients with advanced liver condition "CHILD score ≥ B9"
* Patients with advanced HCC status (BCLC≥ B)
* Patients with combined HBV ,HIV infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2016-03; Primary Completion 2019-02 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants With Sustained Virologic Response 12 Weeks After Treatment | 12 weeks after the last dose of study drugs

SECONDARY OUTCOMES:
Percentage of participants with virologic failure during treatment or relapse after treatment | from baseline until 12 weeks after the last dose of study drugs
Percentage of Participants who will show any radiological or laboratory changes denoting local or denovo recurrence of HCC | Follow up will be done from baseline for up to 36 months for detection of sustained HCC treatment,tumoral progression or denovo occurrence

CONTACTS AND LOCATIONS:
Overall Officials: Gamal Esmat, MD., Principal Investigator — Cairo University; Aisha El Sharkawy, MD, Study Director — Cairo University; Mohamed Hassany, MD, Study Director — National Hepatology & Tropical Medicine Research Institute (NHTMRI); Mai Mehrez, MD., Study Director — National Hepatology & Tropical Medicine Research Institute (NHTMRI); Amr Maged, Study Chair — National Hepatology & Tropical Medicine Research Institute (NHTMRI)
Locations (1):
- Amr Maged, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hassany M, Elsharkawy A, Maged A, Mehrez M, Asem N, Gomaa A, Mostafa Z, Abbas B, Soliman M, Esmat G. Hepatitis C virus treatment by direct-acting antivirals in successfully treated hepatocellular carcinoma and possible mutual impact. Eur J Gastroenterol Hepatol. 2018 Aug;30(8):876-881. doi: 10.1097/MEG.0000000000001152. PMID 29727383
- Available data/document: Informed Consent Form — http://www.megafileupload.com/f3sT/Attachments_201656.zip